CLINICAL TRIAL: NCT03143634
Title: The Modular Protocol for Mental Health (MPMH): A Pilot Randomised Clinical Trial of a Transdiagnostic Psychological Treatment for Mood and Anxiety Disorders in Adults
Brief Title: The Modular Protocol for Mental Health (MPMH)
Acronym: MPMH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Collaborators: Cambridgeshire and Peterborough NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP:MH RfPB PB-PG-0214-33072
Record Dates: First submitted 2017-04-27; First posted 2017-05-08 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder; Posttraumatic Stress Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder; Illness Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic; Phobia, Social; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder | interventions — Mental Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor will be masked, as this is a psychological intervention it is not possible to mask the participant, care provider or investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Modular Protocol for Mental Health (Experimental): The Modular Protocol for Mental Health (Psychological Therapy) will last up to 18 regular weekly face-to-face sessions. Treatment follows a standard structured treatment session as per Cognitive Behavioural Therapy. The MPMH Treatment Manual was written by clinical psychologists. The selection and ordering of the modules for treatment will be delivered and determined by the Trial Clinical Psychologist in collaboration with the service-user. The treatment modules include:
  M1. Getting Acquainted M2. Understanding Emotions M3. Managing and Tolerating Emotions M4. Behavioural activation M5. Tackling Avoidance M6. Tackling Unhelpful Thoughts M7. Tackling Unhelpful Habits M8. Overcoming Repetitive Thinking M9. Managing Upsetting Memories and Images M10. Relapse Prevention and Future Orientation
  Interventions: Behavioral: The Modular Protocol for Mental Health
- Treatment-as-usual (Placebo Comparator): For Treatment-as-usual (Psychological Therapy), clinicians will be asked to provide whatever treatment they deem appropriate, including psychological services, medication and referral to other services. TAU will be delivered by high-intensity therapists or clinical psychologists.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: The Modular Protocol for Mental Health — This intervention is based on evidence-based cognitive-behavioural approaches to psychological disorders and offers a flexible approach to treatment delivery that targets the maladaptive processes common to mood and anxiety disorders.
  Arms: The Modular Protocol for Mental Health
Behavioral: Treatment-as-usual — This intervention will consist of psychological therapies delivered by high-intensity therapists or clinical psychologists.
  Arms: Treatment-as-usual

SUMMARY:
Currently, our best psychological treatments for anxiety and mood disorders only focus on individual diagnoses. So, there are separate treatments for Panic Disorder, or Depressive Disorder, or Social Anxiety, etc. These 'diagnosis-specific' treatments work well for people whose problems fit neatly into a single diagnosis. However, they work far less well for people with complex problems involving multiple diagnoses, and 50% of patients fail to respond well to these existing treatments.

The purpose of this study is to test a new psychological treatment for anxiety and mood problems (the Modular Protocol for Mental Health [MPMH]). Instead of focusing on any single diagnosis, MPMH combines the best treatment techniques into 10 modules to target problems common across all of the different mood and anxiety diagnoses (e.g., intense emotions, negative thinking, upsetting memories, distressing habits). MPMH should therefore be a better treatment for the large numbers of individuals whose problems do not fit neatly into a single diagnosis and for whom any treatments targeting a single diagnosis would leave significant difficulties unaddressed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of a unipolar mood, anxiety, stress or obsessive-compulsive disorder with at least one additional comorbid diagnosis according to the DSM-5. The criteria for diagnosis will be based on the Structured Clinical Interview for the DSM (SCID) which assesses disorders according to DSM-5 diagnostic criteria.
* To be eligible participants will also need to score >10 on either the Patient Health Questionnaire (PHQ-9) or Generalised Anxiety Disorder -7 item scale, GAD-7 (see Study Measures above).

Exclusion Criteria:

* Current/past psychosis or bipolar disorder
* Current full diagnosis of substance use disorder
* Organic brain damage
* Complex trauma history or recurrent self-injury requiring specialist services (as deemed by the NHS Clinical Care team)
* Current suicidality that warrants immediate clinical attention and constitutes a current risk of harm to the individual.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Depression symptoms | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Patient Health Questionnaire - 9-item version (PHQ-9; Kroenke & Spitzer, 2002)
Change in Anxiety symptoms | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  General Anxiety Disorder Questionnaire - 7-item version (GAD-7; Spitzer, Kroenke, Williams, & Lowe, 2006)
Change in Level of disability and functional impairment | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Work and Social Adjustment Scale (WSAS; Mundt, J.C. et al., 2002)

SECONDARY OUTCOMES:
Change in symptoms of social phobia, agoraphobia and specific phobia | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  IAPT Phobia Scales (Department of Health/IAPT, 2011). This measure will only be completed by participants with symptoms of social phobia, agoraphobia or specific phobia.
Change in symptoms of social anxiety | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Social Phobia Inventory (SPIN; Connor, Davidson, Churchill, Sherwood, Foa, & Weisler, 2000). This measure will only be completed by participants with symptoms of social anxiety.
Change in symptoms of generalised anxiety | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990). This measure will only be completed by participants with symptoms of generalised anxiety disorder.
Change in symptoms of obsessive-compulsive disorder | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Obsessive-Compulsive Inventory (OCI; Foa, Kozak, Salkovskis, Coles, & Amir, 1998). This measure will only be completed by participants with symptoms of obsessive-compulsive disorder.
Change in symptoms of post-traumatic stress disorder | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Revised Impact of Event Scale (IES-R; Weiss, 2007). This measure will only be completed by participants with symptoms of PTSD.
Change in symptoms of agoraphobia | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Agoraphobia-Mobility Inventory (MI; Chambless, Caputo, Jasin, Gracely, & Williams, 1985). This measure will only be completed by participants with symptoms of agoraphobia.
Change in symptoms of specific phobias | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Fear Questionnaire (FQ; Marks & Mathews, 1979). This measure will only be completed by participants with symptoms of specific phobia.
Change in symptoms of panic disorder | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Panic Disorder Severity Scale - self report version (PDSS-SR; Shear, Brown, Barlow, Money, Sholomskas, Woods, Gorman, & Papp, 1997). This measure will only be completed by participants with symptoms of panic disorder.
Change in symptoms of illness anxiety | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Health Anxiety Inventory - short version (SHAI; Salkovskis, Rimes, Warwick, & Clark, 2002). This measure will only be completed by participants with symptoms of illness anxiety.
Change in level of disability and functional impairment | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Sheehan Disability Scale (SDS; Sheehan, 1983)
Change in expectancy about treatment outcome, as well as the credibility of the treatment | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  The Treatment Credibility / Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000)
Change in ability to contextualize negative events within a wider frame of reference | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski, Kraaij & Spinhoven, 2000)
Change in disengagement from and acceptance of troublesome mental content, rumination | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Experiences Questionnaire (EQ; Fresco et al., 2007)
Intensity with which participants experience 36 different emotions on a typical day | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Differential Emotions Scale (DES; Izard, 1993)
Change in personality functioning on four subscales: Identity, Self-Direction, Empathy, and Intimacy | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Levels of Personality Functioning Scale (LPFS; Morey et al., 2017)
Change in use of NHS services, other mental health services or activities, help at home, and time off work/lost income | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  Healthlines Resource Use Questionnaire (Salisbury, O'Cathain, Edwards, Thomas, Gaunt, Hollinghurst, et al., 2016)
Change in quality of life assessment of health and wellbeing, daily functioning, and general life satisfaction across multiple domains | Baseline (within two weeks of first treatment session), within one week of the final treatment session, three-months following final treatment session
  World Health Organisation (WHO) Quality of Life Inventory (WHOQOL; World Health Organisation, 1998)

OTHER OUTCOMES:
Change in measure of memory specificity | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  Autobiographical Memory Test (Williams & Broadbent, 1986).
Change in cognitive flexibility for emotional information | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  Affective Card Sorting Task (Barcelo, 2003; Deveney & Deldin, 2006)
Change in immediate recall and working memory for neutral information | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  Digit Span Task (Wechsler, 2008)
Change in brief measure of premorbid intelligence | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  National Adult Reading Test (Nelson & Wilson, 1991)
Change in emotional structure (awareness and differentiation) | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  Levels of Emotional Awareness Scale (Lane et al., 1990)
Change in potential neurobiomarkers that may account for risk of disorders and/or predict treatment response (optional component of participation) | Baseline (within two weeks of first treatment session), within one week of the final treatment session
  Functional connectivity during resting state MRI
Change in levels of rumination | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Ruminative Responses Scale of the Response Styles Questionnaire (RRS; Treynor, Gonzalez, Nolen-Hoeksema, 2003)
Change in ability to tolerate distress | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Distress Tolerance Scale (DTS; Simons & Gaher, 2005)
Change in ability to label, perceive, and regulate emotions | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Difficulties with Emotion Regulation Scale (DERS; Gratz & Roemer, 2004)
Change in negative beliefs, thoughts and assumptions | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Dysfunctional Attitudes Scale (DAS; Weissman, 1979)
Change in mindful awareness | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Kentucky Inventory of Mindfulness Skills (KIMS; Baer, Smith, & Allen, 2004)
Change in fear of physical anxiety sensations | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Anxiety Sensitivity Index (ASI; Reiss, Peterson, Gursky, & McNally 1986)
Change in trauma-related beliefs and maladaptive appraisals of intrusive symptoms | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Posttraumatic cognitions inventory - short version (PTCI; Foa, Ehlers, Clark, Tolin, Orsillo, 1999)
Change in implementation of cognitive therapy skills | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  Skills of Cognitive Therapy (SoCT; Jarrett, 2010)
Change in avoidance of internal experiences including thoughts, feelings, physical sensations. | Within one-week pre-delivery of relevant treatment module; within one-week post-delivery of relevant treatment module (varied time-frame)
  The Multidimensional Experiential Avoidance Questionnaire (Gamez, Chmielewski, Kotov, Ruggero, & Watson, 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dalgleish, PhD, Principal Investigator — Medical Research Council Cognition and Brain Sciences Unit
Locations (1):
- MRC Cognition and Brain Sciences Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL: Structured Clinical Interview for DSM-5-Research Version (SCID-5 for DSM-5, Research Version; SCID-5-RV). Arlington, VA, American Psychiatric Association, 2015
- [Background] Newby JM, McKinnon A, Kuyken W, Gilbody S, Dalgleish T. Systematic review and meta-analysis of transdiagnostic psychological treatments for anxiety and depressive disorders in adulthood. Clin Psychol Rev. 2015 Aug;40:91-110. doi: 10.1016/j.cpr.2015.06.002. Epub 2015 Jun 6. PMID 26094079
- [Background] Kroenke, K.; Spitzer, R.L.The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals, Vol 32(9), Sep 2002, 509-515. http://dx.doi.org/10.3928/0048-5713-20020901-06
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] IAPT/Department of Health, The IAPT data handbook version 2.0.1. 2011: Published to Department of Health Website, in electronic PDF format only
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Foa, E.B., Kozak, M.J., Salkovskis, P.M., Coles, M.E., and Amir, N. (1998). The validation of a new obsessive-compulsive disorder scale: The Obsessive-Compulsive Inventory. Psychological Assessment, 10(3), 206-214.
- [Background] Weiss, D.S., The Impact of Event Scale: Revised, in Cross-cultural assessment of psychological trauma and PTSD, J.P. Wilson and C.S. Tang, Editors. 2007, Springer: New York. p. 219-238.
- [Background] Chambless DL, Caputo GC, Jasin SE, Gracely EJ, Williams C. The Mobility Inventory for Agoraphobia. Behav Res Ther. 1985;23(1):35-44. doi: 10.1016/0005-7967(85)90140-8. No abstract available. PMID 3985915
- [Background] Marks IM, Mathews AM. Brief standard self-rating for phobic patients. Behav Res Ther. 1979;17(3):263-7. doi: 10.1016/0005-7967(79)90041-x. No abstract available. PMID 526242
- [Background] Shear MK, Brown TA, Barlow DH, Money R, Sholomskas DE, Woods SW, Gorman JM, Papp LA. Multicenter collaborative panic disorder severity scale. Am J Psychiatry. 1997 Nov;154(11):1571-5. doi: 10.1176/ajp.154.11.1571. PMID 9356566
- [Background] Salkovskis PM, Rimes KA, Warwick HM, Clark DM. The Health Anxiety Inventory: development and validation of scales for the measurement of health anxiety and hypochondriasis. Psychol Med. 2002 Jul;32(5):843-53. doi: 10.1017/s0033291702005822. PMID 12171378
- [Background] Sheehan, D.V., The Anxiety Disease. 1983, New York: Charles Scribner and Sons.
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Garnefski N, Rieffe C, Jellesma F, Terwogt MM, Kraaij V. Cognitive emotion regulation strategies and emotional problems in 9 - 11-year-old children: the development of an instrument. Eur Child Adolesc Psychiatry. 2007 Feb;16(1):1-9. doi: 10.1007/s00787-006-0562-3. Epub 2006 Jun 21. PMID 16791542
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Izard CE, Libero DZ, Putnam P, Haynes OM. Stability of emotion experiences and their relations to traits of personality. J Pers Soc Psychol. 1993 May;64(5):847-60. doi: 10.1037//0022-3514.64.5.847. PMID 8505713
- [Background] Morey LC. Development and initial evaluation of a self-report form of the DSM-5 Level of Personality Functioning Scale. Psychol Assess. 2017 Oct;29(10):1302-1308. doi: 10.1037/pas0000450. Epub 2017 Feb 27. PMID 28240933
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Salisbury C, O'Cathain A, Edwards L, Thomas C, Gaunt D, Hollinghurst S, Nicholl J, Large S, Yardley L, Lewis G, Foster A, Garner K, Horspool K, Man MS, Rogers A, Pope C, Dixon P, Montgomery AA. Effectiveness of an integrated telehealth service for patients with depression: a pragmatic randomised controlled trial of a complex intervention. Lancet Psychiatry. 2016 Jun;3(6):515-25. doi: 10.1016/S2215-0366(16)00083-3. Epub 2016 Apr 27. PMID 27132075
- [Background] Treynor, W., R. Gonzalez, and S. Nolen-Hoeksema, Rumination Reconsidered: A Psychometric Analysis. Cognitive Therapy and Research 2003. 27(3): p. 247-259.
- [Background] Simons, J.S. and R.M. Gaher, The Distress Tolerance Scale: Development and Validation of a Self-Report Measure. Motivation and Emotion, 2005. 29(2): p. 83-102.
- [Background] Gratz, K.L. & Roemer, L. Journal of Psychopathology and Behavioral Assessment (2004) 26: 41. doi:10.1023/B:JOBA.0000007455.08539.94
- [Background] Weissman, A.N., The Dysfunctional Attitude Scale: A Validation Study. 1979, University of Pennsylvania.
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875
- [Background] Reiss S, Peterson RA, Gursky DM, McNally RJ. Anxiety sensitivity, anxiety frequency and the prediction of fearfulness. Behav Res Ther. 1986;24(1):1-8. doi: 10.1016/0005-7967(86)90143-9. No abstract available. PMID 3947307
- [Background] Foa, E.B., Ehlers, A., Clark, D.M., Tolin, D.F., Orsillo, S.M., The Posttraumatic Cognitions Inventory (PTCI): Development and validation. Psychological Assessment, 1999. 11(3): p. 303-314.
- [Background] Jarrett RB, Vittengl JR, Clark LA, Thase ME. Skills of Cognitive Therapy (SoCT): a new measure of patients' comprehension and use. Psychol Assess. 2011 Sep;23(3):578-86. doi: 10.1037/a0022485. PMID 21319902
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Watson D. Development of a measure of experiential avoidance: the Multidimensional Experiential Avoidance Questionnaire. Psychol Assess. 2011 Sep;23(3):692-713. doi: 10.1037/a0023242. PMID 21534697
- [Background] Williams JM, Broadbent K. Autobiographical memory in suicide attempters. J Abnorm Psychol. 1986 May;95(2):144-9. doi: 10.1037//0021-843x.95.2.144. No abstract available. PMID 3711438
- [Background] Deveney CM, Deldin PJ. A preliminary investigation of cognitive flexibility for emotional information in major depressive disorder and non-psychiatric controls. Emotion. 2006 Aug;6(3):429-437. doi: 10.1037/1528-3542.6.3.429. PMID 16938084
- [Background] Barcelo F. The Madrid card sorting test (MCST): a task switching paradigm to study executive attention with event-related potentials. Brain Res Brain Res Protoc. 2003 Mar;11(1):27-37. doi: 10.1016/s1385-299x(03)00013-8. PMID 12697260
- [Background] Wechsler, D. (2008). Wechsler Adult Intelligence Scale-Fourth Edition. San Antonio, TX: Pearson.
- [Background] Nelson HE, Wilson J (1991) National Adult Reading Test (NART), NFER-Nelson, Windsor, UK.
- [Background] Lane RD, Quinlan DM, Schwartz GE, Walker PA, Zeitlin SB. The Levels of Emotional Awareness Scale: a cognitive-developmental measure of emotion. J Pers Assess. 1990 Fall;55(1-2):124-34. doi: 10.1080/00223891.1990.9674052. PMID 2231235
- [Derived] Black M, Hitchcock C, Bevan A, O Leary C, Clarke J, Elliott R, Watson P, LaFortune L, Rae S, Gilbody S, Kuyken W, Johnston D, Newby JM, Dalgleish T. The HARMONIC trial: study protocol for a randomised controlled feasibility trial of Shaping Healthy Minds-a modular transdiagnostic intervention for mood, stressor-related and anxiety disorders in adults. BMJ Open. 2018 Aug 5;8(8):e024546. doi: 10.1136/bmjopen-2018-024546. PMID 30082367